CLINICAL TRIAL: NCT04459403
Title: Psychiatric Disturbances in Patients Infected With COVID-19: A Cross Sectional Study
Brief Title: Psychiatric Disturbances and COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government); National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Hend Ibrahim Shousha, Assistant Professor, Cairo University
Other Study IDs: 15-2020/1
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; Psychiatric disturbances; Egypt
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
This observational study aims at Assessment of the prevalence and types Psychiatric disturbances that affects patients with COVID-19 infection with and without previous psychiatric diseases. in addition to, Assessment of the types of Psychiatric disturbances in patients with COVID-19 infection in correlation to age, disease severity, co-morbid conditions and treatments applied

DETAILED DESCRIPTION:
International outbreak of the novel coronavirus (2019- nCoV) raised intense attention of specialists worldwide, including psychiatrists. The five stages of shock-denial, anger, bargaining, depression, and acceptance are experienced by many patients. Coronaphobia is a novel term referring to excessive fear of being infected by coronavirus. The current pandemic necessitates research in different areas of psychiatry, including psychosocial and pharmacological interventions to find evidence-based ways of treatment.

This is a multi-center observational cross-sectional study with consecutive sample that will include patients quarantined due to COVID-19 infection. Adult Patients will be recruited consecutively (convenient sample). Data will be collected from patients in the form of:

Demographic data e.g. Age, Gender, Smoking history, exposure to source transmission Co-morbidities e.g. underlying chronic liver, lung, cardiac or kidney diseases, diabetes mellitus, hypertension Severity of COVID-19 infection: mild, moderate or severe

Psychiatric assessment of patients:

Patients will be subjected to the following questionnaires:

1. The General Health Questionnaire (GHQ-12), Arabic version:

   It is the most extensively used screening instrument for common mental disorders, in addition to being a more general measure of psychiatric well-being. It asks whether the respondent has experienced a particular symptom or behavior recently. Each item is rated on a four-point scale (less than usual, no more than usual, rather more than usual, or much more than usual); it gives a total score of 36 based on the Likert scoring styles (0-1-2-3). It is a brief, simple, easy to complete, and its application in research settings as a screening tool is well documented. GHQ-12 is a consistent and reliable instrument when used in general population samples.
2. Taylor Manifest Anxiety Scale , Arabic version:

   A person answers by reflecting on themselves, in order to determine their anxiety level. It is used to separate normal participants from those who would be considered to have pathological anxiety levels. It consists of 50 true or false questions. It has been proven reliable using test-retest reliability. O'Connor, Lorr, and Stafford found there were five general factors in the scale: chronic anxiety or worry, increased physiological reactivity, sleep disturbances associated with inner strain, sense of personal inadequacy, and motor tension .
3. Beck Depression Inventory (BDI) , Arabic version:

   It is a self-report scale designed to assess symptoms of depression such as sadness, guilt, loss of interest, social withdrawal, increase and decrease in appetite or sleep, suicidal ideation, and other behavioral manifestations of depression over the previous 2 weeks. It can also be used over time to monitor symptoms and to assess response to therapeutic interventions. The inventory is composed of 21 groups of statements on a four-point scale with the patient selecting the one that best matches his or her current state.
4. The Brief-COPE scale , Arabic version :

It is an abbreviated version of the COPE (Coping Orientation to Problems Experienced) Inventory. It is a self-report questionnaire developed to assess a broad range of coping responses. It is one of the best validated and most frequently used measures of coping strategies. The instrument consists of 28 items that measure 14 factors of 2 items each, which correspond to a Likert scale ranged from 0 - 3.

from each center included in this study there is a person responsible for checking completeness of the collected questionnaires

Statistical Analysis Results will be evaluated statistically by the Statistical Package for the Social Sciences (SPSS) version 20 (IBM, 2011). Normality of data will be tested by Kolmogorov-Smirnov test. To describe the data, frequency (percent) and mean± SD will be used. T-test and Pearson correlation test will be used for comparisons and correlations respectively for normally distributed data. Mann-Whitney U test and Spearman correlation test will be used for comparisons and correlations respectively for non-normally distributed data. P-values less than 0.05 will be considered statistically significant and 95 % Confidence interval (CI) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases with COVID-19 defined as a positive result to real-time reverse-transcriptase polymerase-chain-reaction (RT-PCR) assay for nasal and pharyngeal swab specimens

Exclusion Criteria:

* Patients who refuse to be included in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 infection by real time PCR quarantined at isolation hospitals of the Egyptian Ministry of health and population
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Psychiatric well-being, level of anxiety, symptoms of depression and coping strategies questionnaire | 3 months
  The General Health Questionnaire: To measure psychiatric well-being. Taylor Manifest Anxiety Scale: To determine the level of anxiety. Beck Depression Inventory: To assess symptoms of depression. The Brief-COPE scale: To assess coping responses. These questionnaires are combined in one questionnaire filled by the patients. it needs from 15-20 minutes.
Prevalence and types of Psychiatric disturbances in patients with COVID-19 infection | 3 months
  prevalence of each type and correlation with age, disease severity, co-morbid conditions and treatments applied

CONTACTS AND LOCATIONS:
Overall Officials: Hend I Shousha, M.D, Principal Investigator — Cairo University
Locations (3):
- Egypt (3):
  - 15 Mayo Smart Hospital, Cairo
  - National hepatology and tropical medicine research institute, Cairo
  - Students hospital, Giza

REFERENCES:
- [Background] Asmundson GJG, Taylor S. Coronaphobia: Fear and the 2019-nCoV outbreak. J Anxiety Disord. 2020 Mar;70:102196. doi: 10.1016/j.janxdis.2020.102196. Epub 2020 Feb 10. No abstract available. PMID 32078967
- [Background] Huang Y, Zhao N. Generalized anxiety disorder, depressive symptoms and sleep quality during COVID-19 outbreak in China: a web-based cross-sectional survey. Psychiatry Res. 2020 Jun;288:112954. doi: 10.1016/j.psychres.2020.112954. Epub 2020 Apr 12. PMID 32325383
- [Background] Daradkeh TK, Ghubash R, el-Rufaie OE. Reliability, validity, and factor structure of the Arabic version of the 12-item General Health Questionnaire. Psychol Rep. 2001 Aug;89(1):85-94. doi: 10.2466/pr0.2001.89.1.85. PMID 11729557
- [Background] Pevalin DJ. Multiple applications of the GHQ-12 in a general population sample: an investigation of long-term retest effects. Soc Psychiatry Psychiatr Epidemiol. 2000 Nov;35(11):508-12. doi: 10.1007/s001270050272. PMID 11197926
- [Background] TAYLOR JA. A personality scale of manifest anxiety. J Abnorm Psychol. 1953 Apr;48(2):285-90. doi: 10.1037/h0056264. No abstract available. PMID 13052352
- [Background] Fahmi M, Ghali M. Arabic version of Taylor Manifest Anxiety Scale. Egypt Psychiatr 1997; 11:119-126
- [Background] Nawel H, Elisabeth S. Adaptation and validation of the Tunisian version of the Brief COPE Scale. Eur Health Psychol. 2015; 17: 783
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Yoo JH. The Fight against the 2019-nCoV Outbreak: an Arduous March Has Just Begun. J Korean Med Sci. 2020 Feb 3;35(4):e56. doi: 10.3346/jkms.2020.35.e56. No abstract available. PMID 31997618
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Xu J, Zheng Y, Wang M, Zhao J, Zhan Q, Fu M, Wang Q, Xiao J, Cheng Y. Predictors of symptoms of posttraumatic stress in Chinese university students during the 2009 H1N1 influenza pandemic. Med Sci Monit. 2011 Jul;17(7):PH60-4. doi: 10.12659/msm.881836. PMID 21709644